CLINICAL TRIAL: NCT06849076
Title: The Effect of Talocrural Joint Manipulation on Ankle Proprioception in Post-Stroke Patients
Brief Title: The Influence of Talocrural Manipulation on Proprioception in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BEUFTR-6
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Proprioception
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The patients enrolled in the study will receive placebo talocrural joint traction and talocrural joint traction in a randomized sequence. The order of the interventions will be determined by flipping a coin.
Who Masked: Participant, Outcomes Assessor
Masking Description: The evaluator and the researcher administering the intervention will be different. The interventions will be administered to participants randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Talocrural Joint Manipulation Group (Placebo Comparator): In this group, patients will receive placebo talocrural joint manipulation. The application will be similar to that in the experimental group, however, hands will be positioned to avoid creating traction or manipulation force, and this position will be maintained for 20 seconds.
  Interventions: Other: Placebo Talocrural Joint Manipulation
- Talocrural Joint Manipulation Group (Experimental): In this group, talocrural joint manipulation will be applied. After positioning the patient, high velocity low amplitude traction will be applied.
  Interventions: Other: Talocrural Joint Manipulation

INTERVENTIONS:
Other: Placebo Talocrural Joint Manipulation — This intervention is a classic method used to evaluate the effect of talocrural joint manipulation.
  Arms: Placebo Talocrural Joint Manipulation Group
Other: Talocrural Joint Manipulation — This technique, aiming to increase ankle dorsiflexion and mechanoreceptor activation, is based on the application of high velocity low amplitude traction to the joint.
  Arms: Talocrural Joint Manipulation Group

SUMMARY:
The aim of the study is to investigate the effect of talocrural joint manipulation on the ankle proprioception of patients with stroke.

DETAILED DESCRIPTION:
The study, utilizing a randomized crossover design, is planned to be conducted on a minimum of 26 patients with stroke who meet the inclusion and exclusion criteria. Patients included in the study will be randomly assigned to receive both placebo talocrural joint manipulation and talocrural joint manipulation interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Two months or longer elapsed since the stroke,
2. A Mini-Mental State Examination score of 24 or higher,
3. Being between 45 and 75 years of age,
4. Having a Brunnstrom stage of 4 or above

Exclusion Criteria:

1. The presence of severe osteoarthritis in the lower extremity,
2. The presence of cancer or diabetic neuropathy,
3. The presence of vestibular disorder,
4. The presence of lower extremity ulceration or amputation,
5. Hemodynamic instability,
6. The presence of other neurological disorders (such as multiple sclerosis, Parkinson's disease),
7. Having experienced an acute lower extremity injury in the last six weeks,
8. History of lower extremity surgery
9. Lack of available range of motion values required for the ankle proprioception test

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Ankle Proprioception | Change from baseline ankle proprioception immediately after the intervention
  The effect of talocrural joint manipulation on ankle proprioception will be evaluated using the Cybex isokinetic dynamometer. The device will analyze the passive joint position sense of the ankle in various positions.

SECONDARY OUTCOMES:
Ankle Dorsiflexion Measurement | Change from baseline ankle dorsiflexion immediately after the intervention
  For the measurement of dorsiflexion range of motion, patients will be asked to stand facing a wall with the assessed leg positioned at the back. They will place their hands on the wall at shoulder width. While keeping the back knee in at least 20 degrees of flexion and ensuring the foot remains in contact with the ground, they will be instructed to lean forward as far as possible. The dorsiflexion range of motion will then be measured using a spirit level application on an iPhone placed one centimeter above the calcaneal tuberosity.

CONTACTS AND LOCATIONS:
Overall Officials: ömer dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; burak mavuş, M.Sc., Principal Investigator — Bolu Abant İzzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital
Locations (1):
- Bolu İzzet Baysal Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Bolu, Merkez, Turkey (Türkiye)

REFERENCES:
- [Background] Vorkas PA, Shalhoub J, Lewis MR, Spagou K, Want EJ, Nicholson JK, Davies AH, Holmes E. Metabolic Phenotypes of Carotid Atherosclerotic Plaques Relate to Stroke Risk: An Exploratory Study. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):5-10. doi: 10.1016/j.ejvs.2016.01.022. Epub 2016 May 23. PMID 27231199
- [Background] Mansfield A, Inness EL, Mcilroy WE. Stroke. Handb Clin Neurol. 2018;159:205-228. doi: 10.1016/B978-0-444-63916-5.00013-6. PMID 30482315
- [Background] Tyson SF, Hanley M, Chillala J, Selley A, Tallis RC. Balance disability after stroke. Phys Ther. 2006 Jan;86(1):30-8. doi: 10.1093/ptj/86.1.30. PMID 16386060
- [Background] de Haart M, Geurts AC, Huidekoper SC, Fasotti L, van Limbeek J. Recovery of standing balance in postacute stroke patients: a rehabilitation cohort study. Arch Phys Med Rehabil. 2004 Jun;85(6):886-95. doi: 10.1016/j.apmr.2003.05.012. PMID 15179641
- [Background] Mayo NE, Wood-Dauphinee S, Cote R, Durcan L, Carlton J. Activity, participation, and quality of life 6 months poststroke. Arch Phys Med Rehabil. 2002 Aug;83(8):1035-42. doi: 10.1053/apmr.2002.33984. PMID 12161823
- [Background] Li J, Zhong D, Ye J, He M, Liu X, Zheng H, Jin R, Zhang SL. Rehabilitation for balance impairment in patients after stroke: a protocol of a systematic review and network meta-analysis. BMJ Open. 2019 Jul 19;9(7):e026844. doi: 10.1136/bmjopen-2018-026844. PMID 31326927
- [Background] Goto Y, Otaka Y, Suzuki K, Inoue S, Kondo K, Shimizu E. Incidence and circumstances of falls among community-dwelling ambulatory stroke survivors: A prospective study. Geriatr Gerontol Int. 2019 Mar;19(3):240-244. doi: 10.1111/ggi.13594. Epub 2019 Jan 8. PMID 30623545
- [Background] Darekar A, McFadyen BJ, Lamontagne A, Fung J. Efficacy of virtual reality-based intervention on balance and mobility disorders post-stroke: a scoping review. J Neuroeng Rehabil. 2015 May 10;12:46. doi: 10.1186/s12984-015-0035-3. PMID 25957577
- [Background] Liu H, Yin H, Yi Y, Liu C, Li C. Effects of different rehabilitation training on balance function in stroke patients: a systematic review and network meta-analysis. Arch Med Sci. 2023 Jun 21;19(6):1671-1683. doi: 10.5114/aoms/167385. eCollection 2023. PMID 38058731
- [Background] Buvarp D, Rafsten L, Abzhandadze T, Sunnerhagen KS. A cohort study on longitudinal changes in postural balance during the first year after stroke. BMC Neurol. 2022 Aug 30;22(1):324. doi: 10.1186/s12883-022-02851-7. PMID 36042404
- [Background] An M, Shaughnessy M. The effects of exercise-based rehabilitation on balance and gait for stroke patients: a systematic review. J Neurosci Nurs. 2011 Dec;43(6):298-307. doi: 10.1097/JNN.0b013e318234ea24. PMID 22089406
- [Background] Oliveira CB, Medeiros IR, Greters MG, Frota NA, Lucato LT, Scaff M, Conforto AB. Abnormal sensory integration affects balance control in hemiparetic patients within the first year after stroke. Clinics (Sao Paulo). 2011;66(12):2043-8. doi: 10.1590/s1807-59322011001200008. PMID 22189728
- [Background] Powden CJ, Hogan KK, Wikstrom EA, Hoch MC. The Effect of 2 Forms of Talocrural Joint Traction on Dorsiflexion Range of Motion and Postural Control in Those With Chronic Ankle Instability. J Sport Rehabil. 2017 May;26(3):239-244. doi: 10.1123/jsr.2015-0152. Epub 2016 Aug 24. PMID 27632835
- [Background] Marron-Gomez D, Rodriguez-Fernandez AL, Martin-Urrialde JA. The effect of two mobilization techniques on dorsiflexion in people with chronic ankle instability. Phys Ther Sport. 2015 Feb;16(1):10-5. doi: 10.1016/j.ptsp.2014.02.001. Epub 2014 Feb 14. PMID 24679362
- [Background] Pellow JE, Brantingham JW. The efficacy of adjusting the ankle in the treatment of subacute and chronic grade I and grade II ankle inversion sprains. J Manipulative Physiol Ther. 2001 Jan;24(1):17-24. doi: 10.1067/mmt.2001.112015. PMID 11174691
- [Background] Dananberg HJ, Shearstone J, Guillano M. Manipulation method for the treatment of ankle equinus. J Am Podiatr Med Assoc. 2000 Sep;90(8):385-9. doi: 10.7547/87507315-90-8-385. PMID 11021048
- [Background] Fisher BE, Piraino A, Lee YY, Smith JA, Johnson S, Davenport TE, Kulig K. The Effect of Velocity of Joint Mobilization on Corticospinal Excitability in Individuals With a History of Ankle Sprain. J Orthop Sports Phys Ther. 2016 Jul;46(7):562-70. doi: 10.2519/jospt.2016.6602. Epub 2016 Jun 6. PMID 27266885
- [Background] Picelli A, Tamburin S, Cavazza S, Scampoli C, Manca M, Cosma M, Berto G, Vallies G, Roncari L, Melotti C, Santilli V, Smania N. Relationship between ultrasonographic, electromyographic, and clinical parameters in adult stroke patients with spastic equinus: an observational study. Arch Phys Med Rehabil. 2014 Aug;95(8):1564-70. doi: 10.1016/j.apmr.2014.04.011. Epub 2014 May 2. PMID 24792138
- [Background] Cho KH, Lee HJ, Lee WH. Intra- and inter-rater reliabilities of measurement of ultrasound imaging for muscle thickness and pennation angle of tibialis anterior muscle in stroke patients. Top Stroke Rehabil. 2017 Jul;24(5):368-373. doi: 10.1080/10749357.2017.1285745. Epub 2017 Feb 15. PMID 28198659
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Girardi P, Manca M, Gimigliano R, Smania N. Is spastic muscle echo intensity related to the response to botulinum toxin type A in patients with stroke? A cohort study. Arch Phys Med Rehabil. 2012 Jul;93(7):1253-8. doi: 10.1016/j.apmr.2012.02.005. Epub 2012 Apr 12. PMID 22502807
- [Background] Heckmatt JZ, Leeman S, Dubowitz V. Ultrasound imaging in the diagnosis of muscle disease. J Pediatr. 1982 Nov;101(5):656-60. doi: 10.1016/s0022-3476(82)80286-2. PMID 7131136
- [Background] Pillen S, van Keimpema M, Nievelstein RA, Verrips A, van Kruijsbergen-Raijmann W, Zwarts MJ. Skeletal muscle ultrasonography: Visual versus quantitative evaluation. Ultrasound Med Biol. 2006 Sep;32(9):1315-21. doi: 10.1016/j.ultrasmedbio.2006.05.028. PMID 16965971
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Tamburin S, Girardi P, Gimigliano R, Smania N. Accuracy of botulinum toxin type A injection into the gastrocnemius muscle of adults with spastic equinus: manual needle placement and electrical stimulation guidance compared using ultrasonography. J Rehabil Med. 2012 May;44(5):450-2. doi: 10.2340/16501977-0970. PMID 22549655
- [Background] Gao F, Grant TH, Roth EJ, Zhang LQ. Changes in passive mechanical properties of the gastrocnemius muscle at the muscle fascicle and joint levels in stroke survivors. Arch Phys Med Rehabil. 2009 May;90(5):819-26. doi: 10.1016/j.apmr.2008.11.004. PMID 19406302
- [Background] Maganaris CN, Baltzopoulos V. Predictability of in vivo changes in pennation angle of human tibialis anterior muscle from rest to maximum isometric dorsiflexion. Eur J Appl Physiol Occup Physiol. 1999 Feb;79(3):294-7. doi: 10.1007/s004210050510. PMID 10048637
- [Background] Manal K, Roberts DP, Buchanan TS. Optimal pennation angle of the primary ankle plantar and dorsiflexors: variations with sex, contraction intensity, and limb. J Appl Biomech. 2006 Nov;22(4):255-63. doi: 10.1123/jab.22.4.255. PMID 17293622
- [Background] Raj IS, Bird SR, Shield AJ. Reliability of ultrasonographic measurement of the architecture of the vastus lateralis and gastrocnemius medialis muscles in older adults. Clin Physiol Funct Imaging. 2012 Jan;32(1):65-70. doi: 10.1111/j.1475-097X.2011.01056.x. Epub 2011 Sep 25. PMID 22152081
- [Background] Fryer GA, Mudge JM, McLaughlin PA. The effect of talocrural joint manipulation on range of motion at the ankle. J Manipulative Physiol Ther. 2002 Jul-Aug;25(6):384-90. doi: 10.1067/mmt.2002.126129. PMID 12183696